CLINICAL TRIAL: NCT00346047
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Determine the Efficacy and Safety of BTDS Compared to Placebo in Subjects With Moderate to Severe Low Back Pain
Brief Title: Comparison of BTDS (Buprenorphine Transdermal System) and Placebo in Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma K.K. (Industry)
Responsible Party: Mutsukuni Kataoka, Mundipharma K.K.
Organization: Mundipharma Pte Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUP3802
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 0 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Experimental)
  Interventions: Drug: Buprenorphine Transdermal System

INTERVENTIONS:
Drug: Placebo — Corresponding placebo is applied for 12weeks
  Arms: 0
Drug: Buprenorphine Transdermal System — Buprenorphine Transdermal System 5, 10 or 20 mg/patch is applied for 12weeks
  Arms: 1

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of BTDS compared to placebo in subjects with moderate to severe low back pain.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy and safety of buprenorphine transdermal system (BTDS) compared to placebo in subjects with moderate to severe low back pain who have a sub-optimal response to their non-opioid analgesic treatment and require opioid analgesics for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 20 years or older.
* Clinical diagnosis of low back pain for 4 weeks or longer with non-malignant pain etiology.

Exclusion Criteria:

* Subjects who have a current chronic disease(s) or who have a past history and high possibilities to relapse, in addition to low back pain, requiring frequent analgesic therapy (e.g. headache, fibromyalgia, gout, rheumatoid arthritis, osteoarthritis and diabetic neuropathy).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The time to the development of inadequate analgesia. | Up to 12weeks

SECONDARY OUTCOMES:
Percentage of subjects who developed inadequate analgesia, 'Average pain over the last 24 hours' scores | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mutsukuni Kataoka, Study Chair — Department Head, Clinical Trial Operations, Clinical Development, Mundipharma K.K.
Locations (29):
- Japan (29):
  - Investigational Site, Ichikawa, Chiba
  - Investigational Site, Matsudo, Chiba
  - Investigational Site, Noda, Chiba
  - Investigational Site, Asakura, Fukuoka
  - Investigational Site, Fukuoka, Fukuoka
  - Investigational Site, Wakasugi, Fukuoka
  - Investigational Site, Takasaki, Gunma
  - Investigational Site, Sapporo, Hokkaido
  - Investigational Site, Kobe, Hyōgo
  - Investigational Site, Yūki, Ibaraki
  - Investigational Site, Kanazawa, Ishikawa-ken
  - Investigational Site, Komatsu, Ishikawa-ken
  - Investigational Site, Hanamaki, Iwate
  - Investigational Site, Morioka, Iwate
  - Investigational Site, Yokohama, Kanagawa
  - Investigational Site, Sendai, Miyagi
  - Investigational Site, Niigata, Niigata
  - Investigational Site, Osaka, Osaka
  - Investigational Site, Yao, Osaka
  - Investigational Site, Koshigaya, Saitama
  - Investigational Site, Tokorozawa, Saitama
  - Investigational Site, Hikone, Shiga
  - Investigational Site, Adachi City, Tokyo
  - Investigational Site, Arakawa City, Tokyo
  - Investigational Site, Edogawa City, Tokyo
  - Investigational Site, Ōta-ku, Tokyo
  - Investigational Site, Suginami, Tokyo
  - Investigational Site, tabashi City, Tokyo
  - Investigational Site, Toshima City, Tokyo